# Analyzing Cervical Cancer Clinical Trials: A Look at the Patterns in Medical Research Participation among Patients with Cervical Cancer

An Informed Consent Form Made For For <u>Power Clinical Trial's</u> Observational Clinical Study

Date: March 16, 2023

#### Preliminaries and Essential Notes

You must give us your consent in order to participate in our study project. Participation in the research is entirely optional, and you are free to do so at any time. This is a quick summary of the study, and this permission form gives more details.

- To find out why a patient enrolls in, stays in, or withdraws from a clinical trial, the study's primary procedures include answering questionnaires and making follow-up calls.
- Given that this is an observational clinical research, the risk to the participants is quite low. If you want to take part, there might not be a clear medical advantage.
- The findings of this study will contribute to our understanding of the factors influencing clinical study enrollment rates, which will be helpful for patients with cervical cancer.
- You won't be deprived of any of your standard benefits, privileges, or rights if you choose not to participate in this trial.

We strongly advise you to carefully read the consent form and to ask any questions you may have before making a decision. Before making a decision, it is also suggested that you speak with your family, close friends, trusted advisors, and/or medical specialists.

# The Objective of the Clinical Trial

The percentages of participants in clinical studies haven't always been perfectly representative of a particular group. This research examines the variables that affect a patient's choice to enroll in, discontinue participation in, or resume participation in a clinical trial for cervical cancer. Additionally, in order to evaluate whether any outcomes are statistically significant, we are seeking to recruit individuals from a range of demographic groups.

### The Process of the Clinical Trial

You have cervical cancer and have been asked to take part in our observational clinical research study because you are presently undergoing therapy or treatment in an interventional trial. In this trial, no therapies or drugs are being tested.

Here is a summary of how we conducted our research:

- Recruitment of Participants: To locate cervical cancer patients who have previously taken part in, withdrew from, or finished a clinical study, our research team will use electronic medical record systems.
- 2. **Informed Consent:** If you decide to take part, our staff will go over the objectives of the study with you and provide you with a consent form to sign. We want to make sure you are aware of the study's goals and your rights as a participant.
- 3. **Data Collection:** Every two weeks, participants will be given a questionnaire asking about their demographics, medical history, and the factors that led them to enroll in, leave the clinical trial early, or complete it. Every three months, the research team will also speak with the participants by phone or video chat to learn more about their experiences participating in the study.
- 4. **Data Analysis:** The study team will examine the data gathered to find out what influences patient enrollment, withdrawal, and clinical trial completion. We'll use statistical analysis to find the relationships between the variables.
- 5. **Dissemination of Results:** The results of the study will be presented at conferences and published in scholarly journals for the benefit of clinical trial

stakeholders. The findings will improve patient recruitment and retention in ongoing clinical studies for cervical cancer.

#### Are There Risks Involved

There may be risks associated with taking part in an observational clinical research for cervical cancer. It is important to remember that there may still be dangers even in the absence of experimental interventions like medication treatments or medical procedures.

These dangers might include the chance of privacy violations, the possibility of going through psychological or emotional hardship because of the study's topic, and the possibility of bad results from any operations performed during the trial.

Before deciding to take part in the clinical study, it is strongly advised to carefully go over the informed consent form and discuss any queries or worries with the research team.

#### Are There Benefits Involved

Patients with cervical cancer may benefit from taking part in observational clinical trials since they expand medical knowledge and may lead to better treatment options in the future.

Throughout the project, patients could also have access to expert care and supervision. The patient may not have a direct medical benefit from the observational study since experimental therapies like drugs or surgery are not included.

Each individual should thoroughly weigh the advantages and drawbacks before deciding whether to take part in a clinical trial based on their unique condition and aspirations. Before selecting a choice, patients are advised to explore their options with their doctor and the study staff.

Instances When My Involvement Will Be Stopped

It is important to note that the researcher or sponsor has the authority to discontinue your participation in the study for a range of reasons, even without your consent. These reasons may include the suspension or termination of the investigation, the elimination, suspension, or withdrawal of funding for the study, or if it is deemed to be in your best interest.

Furthermore, if your health deteriorates, if you become pregnant, if you choose not to proceed with the research after being informed of any modifications that may affect you, or if you fail to adhere to the study's guidelines, your involvement may also be halted.

## Clinical Trials for Cervical Cancer Compared to Other Trials

You should be aware that participation in this research study is entirely optional and that you are free to stop at any moment without incurring any consequences.

Visit clinicaltrials.gov, a website run by the National Institutes of Health (NIH) that offers a comprehensive database of <u>cervical cancer studies</u> from all around the world. You may use the website to limit trials based on a number of search criteria, including area and condition.

On Power's reference page, you may also discover a list of <u>cervical cancer clinical trials</u> that are actively accepting participants.

# Online Research on Clinical Trial Diversity

For those who are interested in learning more about clinical trial diversity, there are several online resources accessible. Here are a few articles you might find interesting if you want to learn more about this subject:

Hsu, William, William Speier, and Ricky K. Taira. "Automated extraction of reported statistical analyses: towards a logical representation of clinical trial literature." In *AMIA*. 2012.

Mason, Su, Mahvash Hussain-Gambles, Brenda Leese, Karl Atkin, and Julia Brown. "Representation of South Asian people in randomised clinical trials: analysis of trials' data." *Bmj* 326, no. 7401 (2003): 1244-1245.

These websites can offer insightful information on the problems with clinical trial diversity and the solutions put forth.

## Privacy

The privacy of the personal information gathered for this project is carefully ensured. We cannot, however, promise that your personal information will always stay private. There may be instances in which it is required by law to be shared. No publications or presentations of the research findings will include your name or any other information that may be used to identify you personally.

Your medical information may be accessed by a number of organizations for the purposes of research, quality assurance, and data analysis, including accrediting bodies, government and regulatory authorities (like the FDA and OHRP), safety monitors, study sponsors, and authorized sponsor representatives.

On rare occasions, we could ask you to fill out an "Authorization Form" outlining how and with whom we might use your information for the study. Before sharing any information or research samples you submitted for this study with other Power researchers, researchers from other university institutions, or researchers from outside commercial firms for upcoming research, we will first get your further informed consent. You can be confident that your private data will be removed and kept secret.

# **Consent Agreement**

You recognize and accept the following:

- You have read and comprehend this informed consent form in its entirety. Before
  making a choice, you are urged to discuss this information with others and seek
  out alternative viewpoints.
- You have gotten satisfactory answers to all of your inquiries concerning the research project and its methodologies, as well as all the information you require to take part in the study.
- You have thought over the benefits, drawbacks, and other options for taking part in the research.
- Your voluntary participation in the research study will not have any impact on your ability to exercise your legal rights.

- Any material updates to the research study that potentially have an impact on your decision to continue participating will be communicated to you.
- This permission form was given to you, and you have the chance to ask any questions you might have.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Investigator's Signature | | |
| I answered any queries the patient and verified that they had freely an | | • |
| Signature of Investigator Who | Received Consent | |
| Name of Investigator | Signature of Investigator | <br>Date |